CLINICAL TRIAL: NCT02153853
Title: Does Obesity Increase the Risk of Conversion and Short Term Complications in Laparoscopic Rectal Surgery?
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Amalie Bøggild, MD, MD, Hvidovre University Hospital
Other Study IDs: BMIandRectalCancer
Record Dates: First submitted 2014-05-29; First posted 2014-06-03 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Rectal Cancer; Obesity
MeSH Terms: conditions — Rectal Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectal cancer: Patients undergoing laparoscopic surgery for rectal cancer at the Department of Gastrointestinal Surgery, Hvidovre Hospital, Copenhagen, Denmark.

SUMMARY:
Obesity is on the rise in the Western population and BMI has been shown to be associated with an increased risk of per- and postoperative complications.

The investigators intend to study a population of more than 300 patients undergoing laparoscopic surgery for rectal cancer.

The investigators main outcome measure will be the conversion rate, and the investigators also intend to study other indications of short term complications, such as peroperative bleeding, infection, re-operation and mortality.

The investigators hypothesise that increased BMI does not increase the risk of conversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer undergoing laparoscopic surgery, Hvidovre Hospital, Denmark.

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with rectal cancer treated with laparoscopic surgery at the Department of Gastrointestinal Surgery, Hvidovre Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2014-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Conversion rate | Day 1
  Amount of patients undergoing conversion from laparoscopic to open surgery.

SECONDARY OUTCOMES:
Peroperative Bleeding | Day 1
  Peroperative blood loss measured in mL.
Length of Hospital Stay | Time of Discharge (3-80 days after surgery, mean: 11 days)
  Days in hospital after surgery.
Short term complications | Time of Discharge (3-80 days after surgery, mean: 11 days)
  Complications at the time of discharge classified according to Clavien Dindo, groups 0-5.
Readmission within 30 days after surgery | 30 days after discharge
  +/- Readmission to the Gastrointestinal Surgical ward within 30 days after initial discharge.
30-day mortality | 30 days after surgery
Duration of surgery | Day 1
  Duration of surgery measured in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Copenhagen, Denmark

REFERENCES:
- See also: Hvidovre Hospital — http://www.hvidovrehospital.dk/menu/